CLINICAL TRIAL: NCT06313125
Title: Comparison of Effects Three-Dimensional Foot-Ankle Exercise and Hip Abductor and External Rotator Strengthening Exercise With Flexible Flatfoot Individuals: Randomized Controlled Study
Brief Title: Comparison of Exercise Effects in Individuals With Flatfoot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Dilek Hande Esen, MSc, PT, Principal Investigator, Toros University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-77082166-302.08.01-796166
Record Dates: First submitted 2024-03-02; First posted 2024-03-15 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Flat Foot [Pes Planus] (Acquired), Unspecified Foot

STUDY DESIGN:
Intervention Model Description: There will be three groups in the study. Short-foot exercise for the control group; short-foot and 3-dimensional foot-ankle exercise for the foot-ankle group; short-foot and clam exercise will be applied for the hip group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The evaluator researcher and participants will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foot-ankle exercise group (Experimental): In the foot-ankle exercise group, three-dimensional foot-ankle extension exercises will be applied in the Proprioceptive Neuromuscular Facilitation (PNF) pattern, in diagonal 1 and 2 directions and short-foot exercise.
  Interventions: Other: 3-dimensional foot-ankle extension exercises; Other: Short-foot exercise
- Hip exercise group (Active Comparator): Clam exercise will be given to this group as a hip abductor and external rotator strengthening exercise. In addition, short-foot exercise will be applied.
  Interventions: Other: Clam exercise; Other: Short-foot exercise
- Control group (Active Comparator): The control group will do only short-foot exercise.
  Interventions: Other: Short-foot exercise

INTERVENTIONS:
Other: 3-dimensional foot-ankle extension exercises — In three-dimensional foot-ankle extension exercises, an elastic band will be used to create resistance to the movement and the intensity/severity of the exercise will be between 13 (somewhat difficult) and 15 (difficult) according to the perceived difficulty level on the Borg scale. Exercises will begin with red (light) tape; Progression will be achieved by moving to a higher level band color [green (medium) and blue (difficult) in that order] every two weeks. Exercises will be performed 3 days a week (2 days supervised, 1 day at home), in 3 sets of 10 repetitions, and a 1-minute rest period will be given between sets to reduce fatigue. Short-foot exercises will be performed in 3 sets of 15 repetitions, with a 45-second rest period between sets, every day a week (2 days/week with a physiotherapist; 5 days/week at home) for 6 weeks.
  Other Names: Short-foot exercise
  Arms: Foot-ankle exercise group
Other: Clam exercise — In three-dimensional foot-ankle extension exercises and clam exercise, an elastic band will be used to create resistance to the movement and the intensity/severity of the exercise will be between 13 (somewhat difficult) and 15 (difficult) according to the perceived difficulty level on the Borg scale. Exercises will begin with red (light) tape; Progression will be achieved by moving to a higher level band color [green (medium) and blue (difficult) in that order] every two weeks. Exercises will be performed 3 days a week (2 days supervised, 1 day at home), in 3 sets of 10 repetitions, and a 1-minute rest period will be given between sets to reduce fatigue. Short-foot exercises will be performed in 3 sets of 15 repetitions, with a 45-second rest period between sets, every day a week (2 days/week with a physiotherapist; 5 days/week at home) for 6 weeks.
  Other Names: Short-foot exercise
  Arms: Hip exercise group
Other: Short-foot exercise — In clam exercise, an elastic band will be used to create resistance to the movement and the intensity/severity of the exercise will be between 13 (somewhat difficult) and 15 (difficult) according to the perceived difficulty level on the Borg scale. Exercises will begin with red (light) tape; Progression will be achieved by moving to a higher level band color [green (medium) and blue (difficult) in that order] every two weeks. Exercises will be performed 3 days a week (2 days supervised, 1 day at home), in 3 sets of 10 repetitions, and a 1-minute rest period will be given between sets to reduce fatigue. Short-foot exercises will be performed in 3 sets of 15 repetitions, with a 45-second rest period between sets, every day a week (2 days/week with a physiotherapist; 5 days/week at home) for 6 weeks.

SUMMARY:
Flexible flatfoot deformity, also known as flexible pes planus, is a common pathological condition characterized by decreased medial longitudinal arch height, eversion of the calcaneus and abduction of the forefoot, especially during loading. Conservative treatments are generally considered as the first step in treatment. In conservative treatments, exercise methods are one of the most frequently used interventions. It has been reported that exercise can improve functional outcomes such as navicular drop, plantar pressure distribution, foot posture, balance, and muscle strength in adults with flexible flatfoot. Although it is known that intrinsic muscle strengthening exercises are a frequently used intervention method in foot pathologies, there is a deficiency in the literature regarding studies investigating the effect of the combination of the most basic foot intrinsic muscle strengthening exercises with different exercise interventions on targeted clinical gains. However, the effect of three-dimensional foot-ankle exercise on flat feet is unknown. Additionally, there are a limited number of studies in the literature investigating the effects of hip abductor and external rotator muscle strength training on foot posture in individuals with flat feet. The aim of this thesis study, planned in the light of this information, is to determine the effects of three-dimensional foot-ankle extension exercises and hip abductor-external rotator muscle strengthening exercise primarily on navicular drop and MLA height in individuals with flexible flat feet; Secondly, it is to examine and compare the effects of static foot posture, hip abductor/external rotator, ankle circumference and intrinsic muscle strength on the functional performance of the lower extremity (endurance, dynamic balance and single leg forward jumping performance). To our knowledge, this study will be the first randomized controlled study to examine and compare the effects of two different exercise interventions that exercise the proximal and distal regions in flatfoot rehabilitation, and the results obtained will contribute to the development of better exercise and treatment programs in this population. In individuals with flat feet, when hip abductor/external rotator strengthening exercises or 3D foot-ankle extension exercises in the PNF pattern are added to short-foot exercise, MLA structure, muscle strength and lower extremity function will be improved more, and when these exercises are combined with short-foot exercise, they are comparable to intrinsic muscle strengthening exercises alone. The investigators hypothesized that it would produce superior clinical results.

DETAILED DESCRIPTION:
This study was designed as an experimental, 3-arm, parallel group, single-blind randomized controlled study that included a 6-week intervention period. The study will be carried out in the university physiotherapy and exercise laboratory. Flat-footed individuals aged between 18-50 years will be included in this study. G-Power (Windows version 3.1.9.7) statistical program was used to determine the number of participants. Sample size calculation was made based on a similar study in the literature that evaluated the amount of navicular drop after foot intrinsic muscle strength training (the primary outcome measure of this study). Type 1 error probability 0.01; The power was accepted as 0.90 and the number of samples was determined as at least 15 people for each group. By adding the 20% loss rate to this number, it was decided that the required number of participants would be 20 people in total for each group. Participants who were confirmed to be included in the study were evaluated by the lead investigator, who was not involved in the evaluations, using Random Allocation Software (version 2.0) in a single block format, 3-dimensional foot-ankle exercise group (foot muscle exercise group, AEG), hip abductor and external rotator strengthening exercise. will be allocated to three different groups: group (hip muscles exercise group, KEG) and control group (CG). The investigator performing the assessments will be blinded to group allocation. Recording of groups' demographic information and assessment of outcome measures will be performed by a secondary investigative physical therapist who is blinded to group information. The principal investigator physiotherapist will be responsible for training the participants to perform the exercises assigned to them, communicating with the participants to monitor exercise performance and exercise compliance, allocating the groups and ensuring blinding. Outcome measurements will be repeated at the start of treatment and at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age range is 18-50 years
* Navicular drop amount is 10 mm or more
* Getting a value of +6 points or above from the Foot Posture Index

Exclusion Criteria:

* Orthopedic and rheumatological diseases of the spinal region and lower extremities
* Surgery history of the spine and lower extremities
* Neurological and systemic disorders
* Describing lower extremity and/or lower back pain in the last 6 months
* Disorders that may affect cognitive and balance (otitis media, visual impairment, etc.)
* Having received any physiotherapy and rehabilitation treatment for flat feet or hips in the last year
* Body mass index being above normal values (18-24.9 kg/m2)
* Having rigid flat feet and hallux rigidus-limitus deformity
* Doing regular sports or exercise

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Medial longitudinal arch height-Navicular Drop Test | 6 weeks
  To detect flatfoot MLA height will be evaluated by the Navicular Drop Test. According to this test result, if the MLA height is between 5-9 mm, the foot is in neutral position; If it is 4 mm or lower, the foot is in supination; If the value is 10 mm or more, a classification can be made as the foot is in pronation. This result will also be used when determining the inclusion criteria, and values of 10 mm and above will be interpreted as low arc.

SECONDARY OUTCOMES:
Static foot posture-Foot Posture Index-6 | 6 weeks
  Static foot posture will be evaluated by the Foot Posture Index-6 survey. While the participant is standing in a comfortable position, first the talus head will be palpated, then the foot will be observed from 3 directions and the remaining items will be evaluated.
Foot structure-Photopodometric analysis | 6 weeks
  Photopodoscopic analysis will be performed with a podoscope device and the Clarke's angle and the Staheli index will be calculated to decide on pronation or supination. The Wejsflog index, hallux valgus angle (ALPHA), and the angle of the varus deformity of the fifth toe (BETA) will be obtained by photophodometer analysis method to detect changes in foot structure. For this, a podoscope (Podo4Foot® CAM) and a special software program (Multireha® software, KOORDYNACJA AS, Radom, Poland) will be used.
Recording demographic and clinical information on the evaluation form | 1 week
  Participants' age (years), gender (female/male), body weight (kg), height (cm), body mass index (kg/m2), dominant side lower extremity (right/left), regular sports habits, injury/surgical history and back or lower extremity complaints will be recorded in the evaluation form prepared by the research administrators. Participants will be asked with which foot they kick the ball, and the foot with which the ball is kicked will be considered the dominant lower extremity.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang C, Chen LY, Liao YH, Masodsai K, Lin YY. Effects of the Short-Foot Exercise on Foot Alignment and Muscle Hypertrophy in Flatfoot Individuals: A Meta-Analysis. Int J Environ Res Public Health. 2022 Sep 22;19(19):11994. doi: 10.3390/ijerph191911994. PMID 36231295
- [Background] Unver B, Erdem EU, Akbas E. Effects of Short-Foot Exercises on Foot Posture, Pain, Disability, and Plantar Pressure in Pes Planus. J Sport Rehabil. 2019 Oct 18;29(4):436-440. doi: 10.1123/jsr.2018-0363. Print 2020 May 1. PMID 30860412
- [Background] Engkananuwat P, Kanlayanaphotporn R. Gluteus medius muscle strengthening exercise effects on medial longitudinal arch height in individuals with flexible flatfoot: a randomized controlled trial. J Exerc Rehabil. 2023 Feb 23;19(1):57-66. doi: 10.12965/jer.2244572.286. eCollection 2023 Feb. PMID 36910682
- [Background] Choi JH, Cynn HS, Yi CH, Yoon TL, Baik SM. Effect of Isometric Hip Abduction on Foot and Ankle Muscle Activity and Medial Longitudinal Arch During Short-Foot Exercise in Individuals With Pes Planus. J Sport Rehabil. 2020 Jul 27;30(3):368-374. doi: 10.1123/jsr.2019-0310. PMID 32717719
- [Derived] Esen DH, Duman T, Tas S, Karatas N. Three-dimensional foot-ankle exercise versus clam exercise in addition to short-foot exercise in individuals with flexible flatfoot: a randomized controlled trial. Physiother Theory Pract. 2025 Oct;41(10):2043-2054. doi: 10.1080/09593985.2025.2492166. Epub 2025 Apr 17. PMID 40244701
- See also: The effects of Dynamic® taping on vertical jumps in adolescent volleyball players with low medial longitudinal arch — https://www.balticsportscience.com/journal/vol14/iss4/4/